CLINICAL TRIAL: NCT01599286
Title: Short-Term Outcome of N-Carbamylglutamate in the Treatment of Acute Hyperammonemia
Acronym: STO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mendel Tuchman (Other)
Collaborators: Children's National Research Institute (Other); Boston Children's Hospital (Other); University Hospitals Cleveland Medical Center (Other); University of California, Los Angeles (Other); Children's Hospital of Philadelphia (Other); Stanford University (Other); Icahn School of Medicine at Mount Sinai (Other); University of Pittsburgh (Other); Children's Hospital Colorado (Other)
Responsible Party: Sponsor-Investigator, Mendel Tuchman, Scientific Director, Children's Research Institute, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCGC0008
Record Dates: First submitted 2012-05-11; First posted 2012-05-16 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-01

CONDITIONS: Propionic Acidemia, Type I and/or Type II; Methylmalonic Acidemia; Carbamoyl-Phosphate Synthase I Deficiency Disease; Ornithine Carbamoyltransferase Deficiency
Keywords: Hyperammonemia; Propionic Acidemia (PA); Methylmalonic Acidemia (MMA); Late-Onset CPS1 Deficiency (CPSD); Late-Onset Ornithine Transcarbamylase Deficiency (OTCD); Carbaglu
MeSH Terms: conditions — Propionic Acidemia; Methylmalonic acidemia; Carbamoyl-Phosphate Synthase I Deficiency Disease; Ornithine Carbamoyltransferase Deficiency Disease; Hyperammonemia | interventions — carglumic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Comparator (Experimental): Parallel Trial Comparing NCG + Standard of Care Treatment
  Interventions: Drug: Carbaglu
- Placebo Comparator (Active Comparator): Placebo and Standard of Care Therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carbaglu — Carbaglu Chemical Composition: N-carbamoyl-L-glutamic acid (NCG)
  The daily dose will be 150 mg/kg/ day or 3.3 g/m2/day for patients >15 kg and will be administered for 7 days or until discharge, whichever is sooner. The doses are to be divided into 2 equal doses and administered orally or enterally by nasogastric or gastrostomy tube. Standard of care will prevail when choosing the mode of drug administration.
  The tablets must be dispersed in a minimum of 2.5-10 ml of water and ingested immediately or administered by fast-push through a syringe via a nasogastric or gastrostomy tube. The suspension has a slightly acidic taste.
  Other Names: Carglumic Acid
  Arms: Active Comparator
Drug: Placebo — Placebo that looks/tastes the same as NCG and is administered on the same schedule as the NCG intervention
  Arms: Placebo Comparator

SUMMARY:
The overall objective of this drug trial is to determine whether the treatment of acute hyperammonemia with N-carbamyl-L-glutamate (NCG, Carglumic acid) in propionic acidemia (PA), methylmalonic acidemia (MMA), late-onset CPS1 deficiency (CPSD) and late-onset Ornithine transcarbamylase deficiency (OTCD) accelerates the resolution of hyperammonemia efficiently and safely.

The primary goal is to determine if the study drug (NCG) efficiently reduces ammonia levels following a hyperammonemia episode(s).

Secondly, the investigators want to know if treatment with this study drug (NCG) efficiently improves neurologic function, reduces plasma glutamine levels and lessens the duration of hospitalization after each episode of hyperammonemia.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized clinical drug trial to evaluate the efficacy of NCG in the treatment of two organic acidemias (severe PA and MMA), and two urea-cycle disorders (late-onset CPSD and OTCD).

Primarily, the investigators want to determine whether NCG treatment of acute hyperammonemia in severe, neonatal-onset PA, MMA, CPSD, and OTCD is efficacious and whether it is safe. The investigators will approach this task in two ways.

1. Assess Whether NCG Treatment is Effective

   The objective of this study is to assess whether NCG is efficacious in treating hyperammonemia and improving outcome:

   The investigators will realize this goal by randomizing each hyperammonemic episode from every subject to NCG (NCG)+standard treatment (NCG-STD) versus placebo+standard treatment (PLBO-STD) and subsequently gauging response with the primary outcome of plasma ammonia levels, in addition to the plasma glutamine, the Functional Status Scale, and the length of hospitalization.
2. Safety

The primary safety outcome of the study will be the assessed via the rate of Serious Adverse Events (SAEs), defined in this study as death or substantial prolongation of hospitalization, as patients are hospitalized as part of the entry to the study.

Safety tests consisting of complete blood count (CBC), liver and kidney function tests, and coagulation profile (PTT/INR) will be performed before treatment, between days 3-5 of treatment, and just prior to discontinuation of NCG. An electrocardiogram will be performed before treatment and on the third day of treatment or before discharge if earlier.

ELIGIBILITY:
Inclusion Criteria

o Aged older than 1 week with an established diagnosis of CPSD or OTCD (as follows):

* Diagnosed with late-onset CPSD confirmed by detection of pathogenic mutation(s), and/or decreased (<20% of control) CPS enzyme activity in liver OR
* Diagnosed with late-onset OTCD by detection of pathogenic OTC mutation, OR decreased (<20% of control) OTC enzyme activity in liver OR elevated urinary orotate (greater than 20 µM/mM) following allopurinol loading with the absence of argininosuccinic acid

AND: Subject or subject's first-degree relative had plasma ammonia level ≥100 μmol/L >1 week of age

OR

o An established diagnosis of PA or MMA (as follows):

- Diagnosed with PA by semi-quantitative urine organic acid analysis, defined as the presence of elevated Methylcitric acid and normal methylmalonic acid levels and no evidence of biotin related disorders in the organic acid analysis

OR

- Diagnosed with MMA by semi-quantitative urine organic acid analysis, defined as an elevation of methylmalonic acid and no evidence of vitamin B12 dependent disorder on plasma amino acid analysis (B12 dependency is defined by documented B12 responsiveness)

AND: Subject or subject's first-degree relative had plasma ammonia level at any time ≥100 μmol/L

* Able to receive medications orally, by nasogastric (NG)-tube or by gastric (G)-tube
* No concomitant illness which would preclude safe participation as judged by the investigator
* If post-menarcheal must have a negative pregnancy test prior to administration of study drug at each episode
* Signed informed consent by the subject or the subject's legally acceptable representative

Exclusion Criteria

* Administration of NCG within 7 days of participation in the study
* Use of any other investigational drug, biologic, or therapy
* Planned participation in any other clinical trial
* Diagnosis of any medical condition causing hyperammonemia which is not PA/MMA, CPSD or OTCD. Other urea cycle disorders will be excluded from this study
* Any clinical or laboratory abnormality or medical condition that, at the discretion of the investigator, may put the subject at additional risk by participating in this study
* Has had a liver transplant
* Is not expected to be compliant with this study in terms of returning to the site for subsequent episodes of hyperammonemia crises
* Is pregnant

Ages: 1 Week to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mendel Tuchman, MD, Principal Investigator — Children's National Research Institute
Locations (9):
- United States (9):
  - University of California Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - The Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital Boston, Boston, Massachusetts
  - Mount Sinai School of Medicine, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
This is a blinded study, the individual participant data will not be shared

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 65 eligible patients, 35 were enrolled with a randomization of hyperammonemia. Eligible patients were randomized at each episode of hyperammonemia. To be enrolled, a patient had to have an eligible episode of hyperammonemia and was then randomized to either placebo or NCG at each randomization. 13 patients had multiple randomizations, 22 only had one.
Units Other Than Participants: Episodes
Groups:
- Episodes of N-Carbamylglutamate: Episodes where the participant was randomized to the NCG arm
- Episodes of Placebo: Episodes where the participant was randomized to the placebo arm
Period: Overall Study
Arm/Group | Episodes of N-Carbamylglutamate | Episodes of Placebo
Started | 24; 54 Episodes | 23; 52 Episodes
Completed | 24; 54 Episodes | 23; 52 Episodes
Not Completed | 0; 0 Episodes | 0; 0 Episodes

BASELINE CHARACTERISTICS:
Population: 65 participants were eligible based on diagnosis. There were 35 individual participants enrolled due to a hyperammonemia episode. 24 individuals had episodes where they were randomized to the NCG arm, and 23 had episodes where they were randomized to the placebo arm. 13 participants had multiple randomizations to both arms throughout the study, while 22 participants only had a single randomization to either placebo of NCG. 35 unique participants were randomized providing 106 randomized episodes.
Units Other Than Participants: Episodes
Groups:
- Episodes of N-carbamylglutamate (NCG): Total number of episodes of hyperammonemia where a patient was randomized to the NCG arm
  A daily dose of 150 mg/kg/ day or 3.3 g/m2/day for patients >15 kg administered for 7 days or until discharge, whichever is sooner.
- Episodes of Placebo: Total number of episodes of hyperammonemia where a patient was randomized to the placebo arm
  Placebo that looks/tastes the same as NCG and is administered on the same schedule as the NCG intervention
- Total: Total of all reporting groups
Arm/Group | Episodes of N-carbamylglutamate (NCG) | Episodes of Placebo | Total
Number analyzed (Participants) | 24 | 23 | 35
Number analyzed (Episodes) | 52 | 54 | 106
Age, Customized [Count of Units; unit: Episodes]
  0 - <5 years | 10 | 16 | 26
  5 - <12 years | 27 | 22 | 49
  12 - <18 years | 1 | 4 | 5
  18+ years | 14 | 12 | 26
Sex: Female, Male [Count of Units; unit: Episodes]
  Female | 33 | 34 | 67
  Male | 19 | 20 | 39
Ethnicity (NIH/OMB) [Count of Units; unit: Episodes]
  Hispanic or Latino | 13 | 17 | 30
  Not Hispanic or Latino | 39 | 36 | 75
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Units; unit: Episodes]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 19 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 11 | 11 | 22
  White | 17 | 19 | 36
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to the Primary Outcome (Earlier of Ammonia <50 µmol/L or Hospital Discharge)
Description: The composite primary intention to treat (ITT) outcome of the earlier of time to reach an ammonia level of ≤50 µmol/L or hospital discharge. Data presented as a hazard ratio based on the time to reach an ammonia level of ≤50 µmol/L. The outcome measure was a survival analysis based on time to reach the earlier of an ammonia level of ≤50 µmol/L or time to discharge, which was considered to be a point where the patient was no longer at risk of neurological injury from ammonia. The outcome of survival analysis was a hazard ratio reflecting the ratio of probabilities in each group (drug vs placebo) of reaching the earlier of an ammonia level of ≤50 µmol/L or discharge. We measured multiple post-treatment ammonia levels at uncontrolled times during an episode, so it is difficult to compute a meaningful average that would not be biased by the frequency and timing of ammonia testing during episodes.
Time Frame: Average of all measurements of hyperammonemia, for up to 7 days
Population: Patients were randomized to either study drug or placebo at each episode of hyperammonemia analysed by diagnosis. Data presented as a hazard ratio based on the time to reach an ammonia level of ≤50 µmol/L. Higher ratios reflect an NCG advantage.
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Units Other Than Participants: Episodes
Groups:
- PA/MMA Episodes: All episodes where a patient diagnosed with PA/MMA was randomized to either placebo or NCG
- CPS1D/OTCD Episodes: All episodes where a patient diagnosed with CPS1D/OTCD was randomized to either placebo or NCGPatients PA/MMA who received study drug
Arm/Group | PA/MMA Episodes | CPS1D/OTCD Episodes
Number analyzed (Participants) | 24 | 11
Number analyzed (Episodes) | 90 | 16
Hazard Ratio | 1.37 [0.88 to 2.13] | 0.79 [0.22 to 2.81]

ADVERSE EVENTS:
Time Frame: During each hospitalization, once per day, up to 7 days.
Description: Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Groups:
- Placebo: Episodes where the patient was randomized to placebo
- N-carbamylglutamate (NCG): Episodes where the patient was randomized to NCG
Arm/Group | Placebo | N-carbamylglutamate (NCG)
All-Cause Mortality (participants affected / at risk) | 10/24 | 14/25
Serious Adverse Events (participants affected / at risk) | 6/24 | 8/25
Other Adverse Events (participants affected / at risk) | 9/24 | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | N-carbamylglutamate (NCG) (N=25)
Gastrointestinal Disorders (Gastrointestinal disorders) | 4 (9) | 5 (7)
Infections and Infestations (Infections and infestations) | 2 (2) | 4 (4)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Metabolic and Nutritional (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Nervous System (Nervous system disorders) | 0 (0) | 3 (4)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | N-carbamylglutamate (NCG) (N=25)
Blood/Lymphatic (Blood and lymphatic system disorders) | 3 (4) | 4 (6)
Cardiac (Cardiac disorders) | 1 (1) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 4 (9) | 4 (8)
General (General disorders) | 3 (5) | 1 (2)
Infections (Infections and infestations) | 3 (4) | 1 (1)
Injury/Procedure Complications (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Investigations (Investigations) | 0 (0) | 3 (6)
Metabolism (Metabolism and nutrition disorders) | 4 (9) | 6 (7)
Nervous System (Nervous system disorders) | 2 (3) | 4 (4)
Product Issues (Product Issues) | 1 (1) | 0 (0)
Psychiatric (Psychiatric disorders) | 0 (0) | 1 (2)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vascular (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT01599286/Prot_SAP_000.pdf